CLINICAL TRIAL: NCT00162890
Title: Evaluation and Physical Therapy for Patients With Degenerated Cervical Spine
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: National Taiwan University, Department and Graduate School of Physical Therapy
Other Study IDs: 9100002264
Record Dates: First submitted 2005-09-12; First posted 2005-09-13 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2009-12

CONDITIONS: Degenerated Cervical Spine; Spinal Diseases
Keywords: degenerated cervical spine; assessment; physical therapy
MeSH Terms: conditions — Spinal Diseases | interventions — Exercise Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patient with degenerative cervical disease
  Interventions: Behavioral: Therapeutic exercise

INTERVENTIONS:
Behavioral: Therapeutic exercise

SUMMARY:
The specific aims are as follows:

1. To investigate the degree of impairment, such as range, proprioception, sensation, and electromyography (EMG) pattern of healthy, older subjects.
2. To investigate the relationship of these impairment measurements, the functional outcome and disability in patients with cervical spondylosis.
3. To develop an exercise program with an emphasis on proprioception, stability and coordination for patients with neck-shoulder complaints to decrease the impairment and increase the functions of patients.

ELIGIBILITY:
Inclusion Criteria:

* Group one: participants without degenerated disease in the cervical spine
* Group two: participants with degenerated disease in the cervical spine

Exclusion Criteria:

* Grade III, IV of degenerated cervical spine

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects aged 20-75 year-old will be recruited. One hundred participants are anticipated to be recruited in this study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2002-02; Primary Completion 2002-07 (Actual); Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shwu-Fen Wang, Ph.D, Study Chair — School and Graduate Institute of Physical Therapy, National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy, National Taiwan University, Taipei, Taiwan